CLINICAL TRIAL: NCT01544179
Title: A Phase III Randomised, Double Blind, Placebo Controlled, Parallel, Multicentre Study to Assess the Efficacy and Safety of Continuing IRESSA 250 mg in Addition to Chemotherapy Versus Chemotherapy Alone in Patients Who Have Epidermal Growth Factor Receptor (EGFR) Mutation Positive Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) and Have Progressed on First Line IRESSA
Brief Title: A Study of IRESSA Treatment Beyond Progression in Addition to Chemotherapy Versus Chemotherapy Alone
Acronym: IMPRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D791LC00001
Record Dates: First submitted 2012-02-15; First posted 2012-03-05 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; Gefitinib; Pemetrexed; Treatment Beyond Progression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gefitinib (Experimental): Gefitinib and cisplatin plus pemetrexed combination chemotherapy
  Interventions: Drug: Gefitinib; Drug: Pemetrexed; Drug: Cisplatin
- Placebo (Placebo Comparator): Placebo and cisplatin plus pemetrexed combination chemotherapy.
  Interventions: Drug: Placebo; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Gefitinib — Investigational Drug
  Arms: Gefitinib
Drug: Placebo — Matching placebo as comparator
  Arms: Placebo
Drug: Pemetrexed — Chemotherapy (concomitant therapy)
Drug: Cisplatin — Chemotherapy (concomitant therapy)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of gefitinib in patients who have progressed on first line gefitinib, comparing continuing gefitinib in addition to cisplatin plus pemetrexed combination chemotherapy versus cisplatin plus pemetrexed combination chemotherapy alone.

DETAILED DESCRIPTION:
A Phase III Randomised, Double blind, Placebo controlled, Parallel, Multicentre Study to Assess the Efficacy and Safety of continuing IRESSA 250 mg in addition to Chemotherapy versus Chemotherapy alone in Patients who have Epidermal Growth Factor Receptor (EGFR) Mutation Positive Locally advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) and have progressed on First Line IRESSA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older (For Japan only- male or female patients aged 20 years or older)
* Cytological or histological confirmation of NSCLC other than predominantly squamous cell histology with an activating EGFR TK mutation as determined locally
* Patients with documented 'acquired resistance' on first line gefitinib
* Patients suitable to start cisplatin based pemetrexed combination chemotherapy.
* Provision of informed consent prior to any study specific procedures.

Exclusion Criteria:

* Prior chemotherapy or other systemic anti-cancer treatment (excluding gefitinib). Palliative bone radiotherapy must be completed at least 2 weeks before start of study treatment with no persistent radiation toxicity).
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease
* Other co-existing malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma or cervical cancer in situ or completely resected intramucosal gastric cancer
* Any evidence of severe of uncontrolled systemic disease Treatment with an investigational drug within 4 weeks before randomization

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2012-03-15 (Actual); Primary Completion 2014-05-05 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Rukazenkov, MD PhD, GCL Oncology, Study Director — AstraZeneca Global R&D, Alderley park, Cheshire, SK10 4TG, UK; Tony Mok, M.D., Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, N.T., Hong KongDepartment of Clinical Oncology, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, N.T., Hong Kong; Jean-Charles Soria, MD, PHD, Principal Investigator — Institute Gustave Roussy, France; Haiyi Jiang, M.D. MSc, Study Director — Zhangjiang Hi-tech Park, 3F, Room 3102, 199 Liangjing Road, Pudong Shanghai, postal code:201203
Locations (48):
- China (16):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chengdu
  - Research Site, Dalian
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Kunming
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
- France (5):
  - Research Site, Clermont-Ferrand
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Villejuif
- Germany (3):
  - Research Site, Hamburg
  - Research Site, Löwenstein
  - Research Site, Würzburg
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Research Site, Budapest, Hungary
- Italy (6):
  - Research Site, Genova
  - Research Site, Parma
  - Research Site, Perugia
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Rozzano
- Japan (5):
  - Research Site, Fukuoka
  - Research Site, Kashiwa
  - Research Site, Sakaishi
  - Research Site, Sayama
  - Research Site, Sunto-gun
- Research Site, Saint Petersburg, Russia
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Zaragoza
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei

REFERENCES:
- [Derived] Soria JC, Wu YL, Nakagawa K, Kim SW, Yang JJ, Ahn MJ, Wang J, Yang JC, Lu Y, Atagi S, Ponce S, Lee DH, Liu Y, Yoh K, Zhou JY, Shi X, Webster A, Jiang H, Mok TS. Gefitinib plus chemotherapy versus placebo plus chemotherapy in EGFR-mutation-positive non-small-cell lung cancer after progression on first-line gefitinib (IMPRESS): a phase 3 randomised trial. Lancet Oncol. 2015 Aug;16(8):990-8. doi: 10.1016/S1470-2045(15)00121-7. Epub 2015 Jul 6. PMID 26159065
- See also: D791LC00001_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=612&filename=D791LC00001_CSR_Synopsis.pdf
- See also: D791LC00001REDACTED_PROTOCOL — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=612&filename=D791LC00001REDACTED_PROTOCOL.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 265 (100%) patients randomised were from 61 centres in 11 countries: 133 patients to the gefitinib group and132 patients to the placebo group. Patients received maximum of 6 cycles cisplatin plus pemetrexed chemotherapy in addition to the randomised treatment (gefitinib or placebo).
Pre-assignment Details: 265 patients were randomised. Randomised patients had epidermal growth factor receptor (EGFR) mutation-positive locally advanced or metastatic non-small cell lung cancer (NSCLC) and who had progressed on first-line gefitinib treatment
Groups:
- Gefitinib: Gefitinib 250mg and cisplatin plus pemetrexed combination chemotherapy
Period: Overall Study
Arm/Group | Gefitinib | Placebo
Started | 133 | 132
Received Treatment | 132 | 132
Did Not Receive Treatment | 1 | 0
Completed | 70 (Patients are ongoing in the study) | 86 (Patients are ongoing in the study)
Not Completed | 63 | 46
Not completed — Death | 50 | 37
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 12 | 7
Not completed — Eligibility criteria not fulfilled | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefitinib | Placebo | Total
Number analyzed (Participants) | 133 | 132 | 265
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 90 | 98 | 188
  >=65 years | 43 | 34 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 84 | 171
  Male | 46 | 48 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 104 | 102 | 206
  Black or African American | 0 | 1 | 1
  White | 29 | 29 | 58

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (Site Read, Investigator Assessment)
Description: PFS is the time from randomisation until the date of objective disease progression as defined by Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) or death (by any cause in the absence of progression). Progression is defined using RECIST (v1.1), as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: Radiologic evaluations were carried out every 6 weeks from randomization until documented progression, withdrawal of consent, loss to follow up, death or the primary data cut off (DCO) for the analysis, assessed up to 50 weeks
Population: Full analysis set (all treated patients)
Measure: Number; unit: Patients with a progression event
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 133 | 132
Patients with a progression event | 98 [4.5 to 5.7] | 107 [4.6 to 5.5]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.273, Cox Proportional Hazards; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.65 to 1.13]

2. Primary Outcome: Median Progression-Free Survival (Site Read, Investigator Assessment)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Full analysis set (all treated patients)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 133 | 132
Months | 5.4 [4.5 to 5.7] | 5.4 [4.6 to 5.5]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from the date of randomisation until death due to any cause. Any subject not known to have died at the time of analysis will be censored based on the last recorded date on which the subject was known to be alive.
Time Frame: Following progression survival data was collected every 8 weeks until documentation of death, withdrawal of consent, loss to follow-up or the final data cut-off, whichever occurs first.
Population: Full analysis set
Measure: Number; unit: Number of patients with an OS event
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 133 | 132
Number of patients with an OS event | 50 [10.4 to 19.0] | 37 [15.6 to NA]

4. Secondary Outcome: Median Overall Survival (OS) at Time of PFS Analysis
Time Frame: Baseline and then every 6 weeks after randomization until objective disease progression. OS is then assessed 8 weekly following PFS progression up to PFS analysis data cut off.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 133 | 132
Months | 14.8 [10.4 to 19.0] | 17.2 [15.6 to NA] — NA because value was Not Calculated, due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.029, Cox Proportional Hazards; Hazard Ratio (HR) = 1.62, 95% CI 2-sided [1.05 to 2.52]

5. Secondary Outcome: Objective Response Rate (ORR) (Site Read Data)
Description: ORR rate is defined as the number (%) of subjects with at least one visit response of Complete Response (CR) or Partial Response (PR) , as defined by Response Evaluation Criteria in Solid Tumours (RECIST v1.1) for target lesions and assessed by CT or MRI. CR, Disappearance of all target lesions; PR, ≥30% decrease in the sum of the longest diameter of target lesions. Data obtained up until progression, or last evaluable assessment in the absence of progression, was included in the assessment of ORR.
Time Frame: Radiologic evaluations were carried out every 6 weeks from randomization until documented progression, withdrawal of consent, loss to follow up, death or the primary data cut off (DCO) for the analysis.
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 133 | 132
Percentage of Participants | 31.6 [0.55 to 1.55] | 34.1 [0.55 to 1.55]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.760, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.55 to 1.55]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is the percentage of patients who achieve disease control at 6 weeks following randomisation. DCR is defined as a Best Objective Response (BOR) of Complete Response, Partial Response or Stable Disease, as defined by Response Evaluation Criteria in Solid Tumours (RECIST v1.1) for target lesions and assessed by CT or MRI. CR, Disappearance of all target lesions; PR, ≥30% decrease in the sum of the longest diameter of target lesions; SD, neither sufficient shrinkage to qualify for PR not sufficient increase to qualify for Progressive Disease (PD); PD, ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, and the sum must have shown an absolute increase of ≥5mm
Time Frame: as for outcome 5
Population: Full analysis set
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 133 | 132
Percentage of Participants | 84.2 [0.74 to 2.62] | 78.8 [0.74 to 2.62]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.308, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.74 to 2.62]

7. Secondary Outcome: Improvement in Trial Outcome Index
Description: An improvement is defined as a change from baseline of ≥ +6 (0-84 score range). Measured by the Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) questionnaire.
Time Frame: At visits 2-8, then every 6 weeks until progression, at progression or treatment discontinuation, and every 8 weeks after progression until PFS analysis data cut off.
Population: Evaluable-for-QoL
Measure: Number; unit: Number of participants improving
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 124 | 129
Number of participants improving | 36 [0.74 to 2.62] | 39 [0.74 to 2.62]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.770, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.53 to 1.59]

8. Secondary Outcome: Time to Worsening in Trial Outcome Index
Description: A worsening is defined as a change from baseline of ≤ -6 (0-84 score range). Measured by the Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) questionnaire
Time Frame: as for outcome 7
Population: Evaluable-for-QoL
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 124 | 129
Weeks | 12.1 [8.7 to 18.1] | 9.4 [7.7 to 13.4]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.507, Cox Proportional Hazards; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.68 to 1.21]

9. Secondary Outcome: Improvement in FACT-L Total Score
Description: An improvement is defined as a change from baseline of ≥ +6 (0-136 score range). Measured by the Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) questionnaire
Time Frame: as for outcome 7
Population: Evaluable-for-QoL
Measure: Number; unit: Number of patients improving
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 124 | 129
Number of patients improving | 44 [0.74 to 2.62] | 49 [0.74 to 2.62]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.725, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.54 to 1.53]

10. Secondary Outcome: Time to Worsening in FACT-L Total Score
Description: A worsening is defined as a change from baseline of ≤ -6 (0-136 score range). Measured by the Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) questionnaire
Time Frame: as for outcome 7
Population: Evaluable-for-QoL
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 124 | 129
Weeks | 12.0 [6.0 to 15.0] | 8.9 [6.0 to 9.9]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.575, Cox Proportional Hazards; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.69 to 1.23]

11. Secondary Outcome: Improvement in Lung Cancer Subscale
Description: An improvement is defined as a change from baseline of ≥ +2 (0-28 score range). Measured by the Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) questionnaire
Time Frame: as for outcome 7
Population: Evaluable-for-QoL
Measure: Number; unit: Number of participants improving
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 124 | 129
Number of participants improving | 54 | 55
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.959, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.61 to 1.68]

12. Secondary Outcome: Time to Worsening in Lung Cancer Subscale
Description: A worsening is defined as a change from baseline of ≤ -2 (0-28 score range). Measured by the Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) questionnaire
Time Frame: as for outcome 7
Population: Evaluable-for-QoL
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Gefitinib | Placebo
Number analyzed (Participants) | 124 | 129
Weeks | 14.6 [9.1 to 24.3] | 9.1 [6.1 to 23.9]
Statistical Analysis 1: Comparison: Gefitinib vs Placebo; Test type: Superiority or Other; p = 0.437, Cox Proportional Hazards; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.66 to 1.20]

ADVERSE EVENTS:
Time Frame: AEs were collected from signature of informed consent, throughout the treatment period until 30 days after discontinuation of the investigational product
Arm/Group | Gefitinib 250 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 38/132 | 28/132
Other Adverse Events (participants affected / at risk) | 125/132 | 129/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib 250 mg (N=132) | Placebo (N=132)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (5) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefitinib 250 mg (N=132) | Placebo (N=132)
Anaemia (Blood and lymphatic system disorders) | 40 (56) | 32 (40)
Bone marrow failure (Blood and lymphatic system disorders) | 4 (7) | 8 (21)
Erythropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Hypercoagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 27 (61) | 22 (53)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 29 (59) | 28 (69)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (11) | 9 (11)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Ichthyosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ototoxicity (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 6 (9) | 4 (6)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1)
Punctate keratitis (Eye disorders) | 0 (0) | 1 (1)
Trichiasis (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 12 (16) | 13 (16)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 34 (58) | 35 (56)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 43 (71) | 19 (22)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 5 (9) | 5 (10)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 4 (6) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 84 (180) | 80 (160)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 14 (15) | 5 (8)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 54 (96) | 43 (75)
Asthenia (General disorders) | 15 (27) | 30 (43)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0)
Face oedema (General disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 28 (37) | 23 (31)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 4 (4) | 2 (2)
Local swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 10 (10) | 9 (15)
Mucosal inflammation (General disorders) | 6 (8) | 3 (4)
Nodule (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 5 (6) | 4 (5)
Pain (General disorders) | 2 (2) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 21 (24) | 14 (15)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1)
Sense of oppression (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 1 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 8 (8)
Cystitis (Infections and infestations) | 6 (6) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (7) | 8 (9)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 6 (6) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Urinary tract infection (Infections and infestations) | 6 (8) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase decreased (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (5) | 11 (17)
Albumin globulin ratio abnormal (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase decreased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 10 (16)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1)
Blood bilirubin decreased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 4 (4)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 12 (14) | 12 (17)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 0 (0)
Blood sodium decreased (Investigations) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 4 (10)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 8 (10) | 4 (5)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 16 (31) | 22 (47)
Occult blood (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 1 (1) | 1 (1)
Palpatory finding abnormal (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 9 (15) | 3 (6)
Protein total decreased (Investigations) | 1 (1) | 0 (0)
Protein urine (Investigations) | 1 (1) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Total bile acids increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 4 (4) | 5 (8)
Weight increased (Investigations) | 3 (8) | 2 (3)
White blood cell count decreased (Investigations) | 17 (38) | 13 (24)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 64 (92) | 45 (74)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemochromatosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (9) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (5)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (9) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (21) | 5 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (9) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (17) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 6 (8) | 3 (4)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 14 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Aphasia (Nervous system disorders) | 2 (2) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Clonic convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9) | 6 (6)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 7 (10)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 11 (14) | 18 (24)
Hypoaesthesia (Nervous system disorders) | 5 (9) | 4 (4)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Mental retardation (Nervous system disorders) | 2 (4) | 3 (8)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 4 (4)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 5 (6) | 7 (8)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (12) | 10 (12)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 2 (2)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 3 (4)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 10 (12) | 7 (7)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 4 (4)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital paraesthesia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (23) | 15 (18)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 9 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 (11) | 7 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 10 (11)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 5 (5)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8 (11) | 4 (4)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (12) | 8 (8)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (9) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 15 (20) | 11 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Erythromelalgia (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 6 (6)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less